CLINICAL TRIAL: NCT04766541
Title: THE ROLE OF CARDIAC MARKERS IN HYPOXIC ISCHEMIC ENCEPHALOPATHY IN LONG-TERM NEURODEVELOPMENTAL FOLLOW UP
Acronym: TRCMHIE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Umit Ayse Tandircioglu, Medical Doctor, Hacettepe University
Other Study IDs: GOHIE
Record Dates: First submitted 2021-02-20; First posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Hypoxic-Ischemic Encephalopathy; Newborn Morbidity
Keywords: newborn; hypoxic ischemic encephalopathy; bayley score; neurodevelopmental follow up
MeSH Terms: conditions — Hypoxia-Ischemia, Brain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — There is no intervention.

SUMMARY:
In this study, the correlation of cardiac marker values (Troponin I, CK, CK-MB) measured before treatment with the long-term neurodevelopmental score of newborns diagnosed with perinatal asphyxia and treated with therapeutic hypothermia with a diagnosis of hypoxic ischemic encephalopathy (HIE) will be evaluated.

Physical examination, laboratory (especially cardiac markers), aEEG findings and diffusion MRI findings of babies who have been hospitalized in the neonatal intensive care unit between 2015-2020 due to respiratory distress and who have undergone perinatal asphyxia but have undergone therapeutic hypothermia treatment will be recorded from their files in the hospital system. The neurological evaluations and neurodevelopmental scores of the babies in the follow-up in the neonatal high risk follow-up clinic after discharge will be recorded from their files.

DETAILED DESCRIPTION:
With therapeutic hypothermia, it is aimed to reduce the temperature of brain structures and basal ganglia to 32- 34 degrees for 72 hours. The mechanism of action of hypothermia can be listed as decrease in cerebral metabolism, inhibition of edema, decrease in energy metabolism, decrease in cytotoxic amino acid and nitric oxide accumulation, inhibition of platelet activating factor and inflammatory cascade, suppression of free radical activity and prevention of cell death.

Perinatal hypoxia not only affects brain tissue, but also all organs. Therefore, the baby's respiratory system, blood gases, cardiac functions and liver functions are evaluated. Electrolyte, blood sugar and blood pressure are closely monitored due to the possibility of adrenal glands being affected. Since gastrointestinal injury is possible, nutrition is done extremely slowly and carefully. The useful markers in determining the neurological prognosis are the neurological findings of the patient as well as the defect in the aEEG monitoring.

Cardiac markers (CK, CK-MB, Troponin-I) have been shown to be a sensitive marker for asphyxia in term infants. Any interruption in the placental blood supply can cause the fetus to undergo hypoxic ischemia with the activation of the 'diving reflex' to protect the most vital organs. However, because myocardial tissue has insufficient reserves to tolerate hypoxia, myocardial injury may occur and an increase in serum troponin I, CK, CK-MB may occur. High levels of cardiac markers are an indicator of ongoing myocardial damage during HIE.

Diffusion MR imaging performed after hypothermia tries to see the damaged areas in the brain. Diffusion MRI and aEEG follow-up have been shown to be prognostic in the literature. Patients with hypothermia are followed up in our neonatal outpatient clinic and monitored in terms of growth and neurodevelopmental aspects.

In this study, the correlation of cardiac marker values (Troponin I, CK, CK-MB) measured before treatment with the long-term neurodevelopmental score of newborns diagnosed with perinatal asphyxia and treated with therapeutic hypothermia with a diagnosis of hypoxic ischemic encephalopathy (HIE) will be evaluated.

Physical examination, laboratory (especially cardiac markers), aEEG findings and diffusion MRI findings of babies who have been hospitalized in the neonatal intensive care unit between 2015-2020 due to respiratory distress and who have undergone perinatal asphyxia but have undergone therapeutic hypothermia treatment will be recorded from their files in the hospital system. The neurological evaluations and neurodevelopmental scores of the babies in the follow-up in the neonatal high risk follow-up clinic after discharge will be recorded from their files.

ELIGIBILITY:
Inclusion Criteria:

* Babies who have been hospitalized in the Neonatal Intensive Care Unit of Hacettepe University İhsan Doğramacı Children's Hospital, have received therapeutic hypothermia treatment for perinatal asphyxia and are discharged and have neurodevelopmental assessments during their follow-up will be taken.

Exclusion Criteria:

* Babies with chromosomal abnormalities Major congenital anomaly (congenital heart disease, lung anomaly, congenital diaphragmatic hernia, spina bifida etc.) Babies with inherited metabolic diseases • Babies with congenital muscle disease-hypotonicity

Max Age: 28 Days | Sex: All
Age Groups: Child
Study Population: Newborns who were born with hypoxic ischemic encephalopathy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Neurodevelopmental follow up Cardiac markers | 12 months
  In this study, the correlation of cardiac marker values (Troponin I, CK, CK-MB) measured before treatment with the long-term neurodevelopmental score of newborns diagnosed with perinatal asphyxia and treated with therapeutic hypothermia with a diagnosis of hypoxic ischemic encephalopathy (HIE) will be evaluated.

SECONDARY OUTCOMES:
Diffusion MRI and cardiac markers correlations | 12 months
  Diffusion MR imaging and correlation with cardiac markers

CONTACTS AND LOCATIONS:
Locations (1):
- Umit Ayse Tandircioglu, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Physical examination, laboratory (especially cardiac markers), aEEG findings and diffusion MRI findings of babies who have been hospitalized in the neonatal intensive care unit between 2018-2020 due to respiratory distress and who have undergone perinatal asphyxia but have undergone therapeutic hypothermia treatment will be recorded from their files in the hospital system. The neurological evaluations and neurodevelopmental scores of the babies in the follow-up in the neonatal high risk follow-up clinic after discharge will be recorded from their files.